CLINICAL TRIAL: NCT03917823
Title: Intercostal Cryoneurolysis Following Traumatic Rib Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Revised protocol to such a significant degree that we simply closed this study and started a new study.
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cryoneurolysis & Rib Fracture
Record Dates: First submitted 2019-04-13; First posted 2019-04-17 (Actual); Results first posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: Rib Fractures
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Intervention Model Description: Randomized, double-masked, sham-controlled, parallel-arm human subjects clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Cryoneurolysis probes are available for a console neurolysis device (PainBlocker, Epimed, Farmers Branch, Texas) that either (1) pass nitrous oxide to the tip inducing freezing temperatures; or, (2) vent the nitrous oxide at the base of the probe so that no gas reaches the probe tip, resulting in no temperature change. The latter is a sham procedure since without the temperature change, no ice ball forms and therefore the target nerve is not affected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cryoneurolysis (active) (Experimental): The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation (active or sham) separated by 1-minute defrost periods.
  Interventions: Device: Cryoneurolysis
- Sham (Sham Comparator): For the sham probes, the nitrous oxide will be vented prior to reaching the probe shaft, resulting in a lack of perineural temperature change.
  Interventions: Device: Sham comparator

INTERVENTIONS:
Device: Cryoneurolysis — The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation separated by 1-minute defrost periods for the target intercostal nerves.
  Arms: Cryoneurolysis (active)
Device: Sham comparator — For the sham probes, the nitrous oxide will be vented prior to reaching the probe shaft, resulting in a lack of perineural temperature change.
  Arms: Sham

SUMMARY:
Rib fractures are one of the most common injuries in trauma patients. These fractures are associated with significant pain as well as decreased ability to inspire deeply or cough to clear secretions, which together lead to pulmonary complications and a high degree of morbidity and mortality. Peripheral nerve blocks as well as epidural blocks have been used with success to improve pain control in rib fracture patients and have been associated with decreased pulmonary complications and improved outcomes. However, a single-injection nerve block lasts less than 24 hours; and, even a continuous nerve block is generally limited to 3-4 days. The pain from rib fractures usually persists for multiple weeks or months. In contrast to local anesthetic-induced nerve blocks, a prolonged block lasting a few weeks/months may be provided by freezing the nerve using a process called "cryoneurolysis". The goal of this randomized, double-masked, sham-controlled study is to evaluate the potential of cryoanalgesia to decrease pain and improve pulmonary mechanics in patients with rib fractures.

DETAILED DESCRIPTION:
Rib fractures represent a significant source of morbidity in trauma patients, with approximately 10% of trauma patients presenting with rib fractures.1 Pain from rib fractures is associated with decreased ability to cough and inspire deeply, predisposing patients to atelectasis and pulmonary complications. Neuraxial blocks, both thoracic epidurals and paravertebral blocks, have been associated not only with decreased pain, but also decreased pulmonary complications and overall mortality in patients with rib fractures.2 Furthermore, intercostal nerve blocks with local anesthetic have been shown to improve pain scores, peak expiratory flow rates, and arterial oxygen saturation on room air.3 However, intercostal nerve blocks are not without risk and incidence of pneumothorax has been reported as 1.4% for each individual intercostal nerve that is blocked.4 Although it is possible that the use of in-plane ultrasound guidance may decrease the risk of pneumothorax, this has not been evaluated. Additionally, intercostal blocks with bupivacaine have been reported to resolve in as little as six hours,5 likely due to the high vascularity and consequent uptake of local anesthetic from the intercostal space.

An alternative analgesic technique is cryoneurolysis, consisting of the application of exceptionally low temperatures to reversibly ablate peripheral nerves, resulting in temporary pain relief termed "cryoanalgesia".6 The intense cold temperature at the probe tip produces Wallerian degeneration-a reversible breakdown of the nerve axon-subsequently inhibiting transmission of afferent and efferent signals. Because the nerve endoneurium, perineurium, and epineurium remain intact, the axon regenerates along the exoskeleton at a rate of approximately 1-2 mm/day. While cryoneurolysis of peripheral nerves through surgical incisions has been commonly used to treat pain since 1961, the development of cryo probes that may be inserted percutaneously promise a revolution in the use of this modality. The combination of newly-designed narrow-gauge probes (upper right) and ultrasound now make percutaneous cryoanalgesia as simple as placing a peripheral nerve block: the probe tip is inserted adjacent to the target nerve under ultrasound guidance, and a series of 2-minute freezing cycles are administered followed by probe withdrawal. The procedure is essentially the same as placing an ultrasound-guided peripheral nerve block; however, instead of injecting local anesthetic, a gas circulates through the probe, inducing cold at the tip and freezing the target nerve. Nothing remains within the patient and there is no external equipment to prepare or manage. Importantly, cryoneurolysis and the probes are already approved by the United States Food and Drug Administration for the treatment of acute and chronic pain, so no additional regulatory approval is required for the proposed clinical trial.

Theoretical benefits of cryoneurolysis include an ultra-long duration of pain control without opioid involvement, no catheter management/removal (reducing infection risk), the lack of an infusion pump and anesthetic reservoir to carry, an extraordinarily-low risk of infection (approaching zero), and no risk of local anesthetic toxicity, catheter dislodgement or leakage. With a single 8-minute percutaneous cryoneurolysis procedure consisting of several freeze/defrost cycles, a truncation of sensory nerve conduction is induced for 6-8 weeks, with the complete restoration of nerve structure and function following remyelination. Cryoneurolysis offers the possibility of potent, side effect-free analgesia outlasting the surgical pain, and obviating the need for postoperative opioids.

All subjects would continue to receive standard and customary analgesics, so there is no risk of subjects receiving a lower degree of analgesia than if they otherwise did not enroll in the study. The cryoneurolysis procedure will be done in addition to the investigator's current UCSD standard practice.

Study Overview

Day 0 Subjects randomized and cryoneurolysis/sham procedure administered

Days 0-4, 7, 14, 21, and Months 1, 3, 6 Data collection

Subjects will be individuals who present to one of the UCSD hospitals with rib fracture(s) and significant pain. Those who consent to participate in this study will have standard intercostal nerve blocks administered.

Treatment group assignment (randomization). Subjects will be allocated to one of two possible treatments:

1. cryoneurolysis
2. sham procedure (placebo control)

Computer-generated randomization lists will be used to create sealed, opaque randomization envelopes with the treatment group assignment enclosed in each envelope labeled with the randomization number.

The specific intercostal nerves targeted will depend on the injury site. The cryoneurolysis sites will be cleansed with chlorhexidine gluconate and isopropyl alcohol. Using the optimal ultrasound transducer for the specific anatomic location and subject anatomy (linear vs curvilinear array), the target nerves will be identified in a transverse cross-sectional (short axis) view.

Cryoneurolysis Procedure: Cryoneurolysis probes are available for a console neurolysis device (PainBlocker, Epimed, Farmers Branch, Texas) that either (1) pass nitrous oxide to the tip inducing freezing temperatures; or, (2) vent the nitrous oxide at the base of the probe so that no gas reaches the probe tip, resulting in no temperature change. The latter is a sham procedure since without the temperature change, no ice ball forms and therefore the target nerve is not affected. An angiocatheter/introducer may be inserted beneath the ultrasound transducer and directed until the probe tip is immediately adjacent to the target nerve (lidocaine 1% will be administered, as needed, to anesthetize the angiocatheter track). The target nerves will be the intercostal nerves above and below each fractured rib. The angiocatheter needle will be removed, leaving the angiocatheter through which the appropriate Epimed probe will be inserted until it is adjacent to the target nerve. The cryoneurolysis device will be triggered using 3 cycles of 2-minute gas activation (active or sham) separated by 1-minute defrost periods. For active probes, the nitrous oxide will be deployed to the tip where a drop in temperature to -70°C will result in cryoneurolysis. For the sham probes, the nitrous oxide will be vented prior to reaching the probe shaft, resulting in a lack of perineural temperature change. The process will be repeated with the same treatment probe for any additional nerves (e.g., all nerves will receive either active cryoneurolysis or sham/placebo, and not a mix of the two possible treatments).

Statistical Analysis: The primary endpoint is average pain score the day following treatment. The primary inference will be based on the Mann-Whitney U test of the difference between groups with an exact test with two-sided Type I error of 5%. Highest spirometry reading for each period of time will be the secondary end point of highest interest [so designated after the 4th subject was enrolled on September 23, 2019].

Patient baseline characteristics will be summarized by group with mean, standard deviation, quartiles, range, and boxplots for continuous data; and counts and percentages for binary and categorical data. Group differences will be assessed with Mann-Whitney U test for continuous data and Pearson chi-square test for categorical data. If any key characteristics are significantly different between groups, a proportional odds model will be used to test for a group difference in the primary outcome adjusting for the potential confounding variable.

Pilot parameters for sample size justification are based on Osinowo et al (2004).3 Of the initial pain scores for n=21 patients, n=18 (86%) had scores of 3.0 and n=3 (14%) had scores of 2.0 (mean 2.86 ± 0.36). After 24 hours n=13 (62%) had scores of 0 and n=8 (38%) had scores of 1.0 (mean 0.38 ± 0.50).

To simulate power with Mann-Whitney U test, we simulate controls groups assuming the distribution of initial average pain scores from Osinowo et al. scores in the cryoneurolysis groups are simulated assuming a score distribution 10% 0, 15% 1, 25% 2, and 50% 3 (resulting in mean 2.12 ± 1.04 compared to control group mean 2.86 ± 0.36).

Under these assumptions a sample size of n=25 per group attains power 84% with two-sided Type I error 5%. To allow for drop-outs, we will enroll up to a maximum of 60 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of at least 18 years of age
* having 1-3 sustained rib fractures on either or both sides (if bilateral fractures, then total up to 6 fractures with up to 3 per side)
* regional anesthetic requested by the admitting service
* accepting of a cryoneurolysis procedure

Exclusion Criteria:

* chronic opioid use (daily use within the 2 weeks prior to surgery and duration of use > 4 weeks
* pregnancy
* incarceration
* inability to communicate with the investigators
* morbid obesity (body mass index > 40 kg/m2)
* possessing any contraindication specific to cryoneurolysis such as a localized infection at the treatment site, cryoglobulinemia, cold urticaria and Reynaud's Syndrome
* any patient unable to correctly perform incentive spirometry as this is an outcome measure
* any patient with any degree of decreased mental capacity as determined by the surgical service
* any reason an investigator believes study participation would not be in the best interest of the potential subject, including an anti-coagulated state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2020-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cryoneurolysis (Active) | Sham
Started | 2 | 2
Completed | 1 | 0
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cryoneurolysis (Active) | Sham | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 59.5 [55 to 64] | 54.5 [43 to 66] | 57.0 [43 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4
Height (m) [Mean (Full Range); unit: meters] | 1.75 [1.7 to 1.8] | 1.75 [1.7 to 1.8] | 1.75 [1.7 to 1.8]
Weight (kg) [Mean (Full Range); unit: kg] | 93.0 [68 to 118] | 97.6 [90.4 to 104.8] | 95.3 [68 to 118]

OUTCOME MEASURES:

1. Primary Outcome: Average Resting Pain Score
Description: Pain score measured using the numeric rating scale for pain: 0=no pain and 10=worst imaginable pain
Time Frame: Day following treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cryoneurolysis (Active) | Sham
Number analyzed (Participants) | 2 | 2
score on a scale | 5.0 (2.8) | 8.3 (1.8)

2. Secondary Outcome: Average Pain Score
Description: Pain score measured using the numeric rating scale for pain: 0=no pain and 10=worst imaginable pain
Time Frame: Days 2-4, Weeks 1-3, Months 1,3,6
Population: One subject from the treatment/experimental group could not be reached Months 3 and 6; one subject from the control group dropped out after postoperative day 1; and one subject from the control group could not be reached Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cryoneurolysis (Active) | Sham
Number analyzed (Participants) | 2 | 2
score on a scale
  Day 2 | 1.5 (2.1) | 8.3 (0.4)
  Day 3: number analyzed (Participants) | 2 | 1
  Day 3 | 3.5 (4.9) | 8.5 (0)
  Day 4: number analyzed (Participants) | 2 | 1
  Day 4 | 1.5 (2.1) | 8.0 (0)
  Week 1: number analyzed (Participants) | 2 | 1
  Week 1 | 2.0 (2.8) | 8.0 (0)
  Week 2: number analyzed (Participants) | 2 | 1
  Week 2 | 1.0 (1.4) | 4.5 (0)
  Week 3: number analyzed (Participants) | 2 | 1
  Week 3 | 1.0 (1.4) | 3.5 (0)
  Week 4: number analyzed (Participants) | 2 | 1
  Week 4 | 1.0 (1.4) | 4.5 (0)
  Month 3: number analyzed (Participants) | 1 | 1
  Month 3 | 1.0 (0) | 3.0 (0)
  Month 6: number analyzed (Participants) | 1 | 0
  Month 6 | 0 (0) |

3. Secondary Outcome: Worst Pain Score
Description: Pain score measured using the numeric rating scale for pain: 0=no pain and 10=worst imaginable pain
Time Frame: Days 1-4, weeks 1-4, months 3 & 6
Population: One patient withdrew and 2 patients were lost to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cryoneurolysis (Active) | Sham
Number analyzed (Participants) | 2 | 2
score on a scale
  Day 1 | 7.5 (3.5) | 9.8 (0.4)
  Day 2 | 4.0 (5.7) | 9.5 (0.7)
  Day 3: number analyzed (Participants) | 2 | 1
  Day 3 | 4.3 (6) | 10
  Day 4: number analyzed (Participants) | 2 | 1
  Day 4 | 3.5 (4.9) | 10
  Week 1: number analyzed (Participants) | 2 | 1
  Week 1 | 3.3 (4.6) | 10
  Week 2: number analyzed (Participants) | 2 | 1
  Week 2 | 3.5 (4.9) | 7.5
  Week 3: number analyzed (Participants) | 2 | 1
  Week 3 | 3.0 (4.2) | 7.0
  Week 4: number analyzed (Participants) | 2 | 1
  Week 4 | 3.0 (4.2) | 5.0
  Month 3: number analyzed (Participants) | 1 | 1
  Month 3 | 4.5 | 7.0
  Month 6: number analyzed (Participants) | 1 | 0
  Month 6 | 0 |

4. Secondary Outcome: Opioid Consumption
Description: Number of opioid tablets consumed previous 24 hours (oxycodone 5 mg)
Time Frame: Days 1-4, 7, 14, 21, and months 1, 3 and 6
Population: One subject withdrew and two subjects were lost to follow-up
Measure: Mean (Standard Deviation); unit: opioid tablets (5mg oxycodone)
Arm/Group | Cryoneurolysis (Active) | Sham
Number analyzed (Participants) | 2 | 2
opioid tablets (5mg oxycodone)
  Day 1 | 5.5 (6.5) | 2.8 (3.9)
  Day 2 | 0.5 (0.7) | 14.5 (4.9)
  Day 3 | 1.0 (1.4) | 18 (10)
  Day 4: number analyzed (Participants) | 2 | 1
  Day 4 | 1.0 (1.4) | 24.0 (0)
  Week 1: number analyzed (Participants) | 2 | 1
  Week 1 | 2.0 (2.8) | 22.0 (0)
  Week 2: number analyzed (Participants) | 2 | 1
  Week 2 | 2.0 (2.8) | 10 (0)
  Week 3: number analyzed (Participants) | 2 | 1
  Week 3 | 1.5 (2.1) | 12.0 (0)
  Week 4: number analyzed (Participants) | 2 | 1
  Week 4 | 0.5 (0.7) | 0 (0)
  Month 3: number analyzed (Participants) | 1 | 1
  Month 3 | 0 (0) | 0 (0)
  Month 6: number analyzed (Participants) | 1 | 0
  Month 6 | 0 (0) |

5. Secondary Outcome: Incentive Spirometer Volume
Description: maximum incentive spirometer volume
Time Frame: Days 1-4, 7, 14, and 21
Population: some subjects were lost to follow-up and one withdrew
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cryoneurolysis (Active) | Sham
Number analyzed (Participants) | 2 | 2
mL
  Day 1 | 2625 (530) | 1675 (1520)
  Day 2 | 2375 (177) | 1575 (1662)
  Day 3: number analyzed (Participants) | 2 | 1
  Day 3 | 2500 (354) | 500
  Day 4: number analyzed (Participants) | 2 | 1
  Day 4 | 2875 (884) | 500
  Day 7: number analyzed (Participants) | 2 | 1
  Day 7 | 2750 (707) | 750
  Day 14: number analyzed (Participants) | 2 | 1
  Day 14 | 2875 (884) | 1250
  Day 21: number analyzed (Participants) | 2 | 1
  Day 21 | 2875 (884) | 1250

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Cryoneurolysis (Active) | Sham
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT03917823/Prot_SAP_001.pdf